CLINICAL TRIAL: NCT06442254
Title: Examining the Effects of Virtual Reality on Early Vital Variables and Spillovers in Intensive Care Patients
Brief Title: The Effects of Virtual Reality in Intensive Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Yasemin Çırak, Principal Investigator, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 23-152
Record Dates: First submitted 2024-05-01; First posted 2024-06-04 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Virtual Reality; Intensive Care Unit Acquired Weakness
Keywords: virtual reality; intensive care; respiratory muscle strength; respiratory function
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Both the participants and the person analyzing the study do not know which is the study and control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): In the intervention group, virtual reality application will be applied in addition to conventional treatment. In the application, which will be done with VR glasses, a video of walking on Istiklal Street in Istanbul's Beyoğlu district will be watched. To evaluate the effectiveness of the application, vital signs, respiratory muscle strength, grip strength, blood gas analysis, dyspnea and fatigue will be evaluated. Additionally, Richmond Agitation Sedation Scale (RASS), Non-Verbal Pain Scale, Glaskow coma scale, Physical Function Test in Intensive Care (PFIT)- CPax (Chelsea Critical Care Physical Assessment Tool) scales will be used.
  Interventions: Other: Virtual Reality
- Control Group (No Intervention): Conventional treatment will be applied in the control group. Participants' vital signs, respiratory muscle strength, grip strength, blood gas analysis, dyspnea and fatigue will be evaluated. Additionally, Richmond Agitation Sedation Scale (RASS), Non-Verbal Pain Scale, Glaskow coma scale, Physical Function Test in Intensive Care (PFIT)- CPax (Chelsea Critical Care Physical Assessment Tool) scales will be used.

INTERVENTIONS:
Other: Virtual Reality — In the application, which will be done with VR glasses, a video of walking on Istiklal Street in Istanbul's Beyoğlu district will be watched.
  Arms: Virtual Reality Group

SUMMARY:
Weakness of respiratory muscles delays weaning from the ventilator, prolongs hospital stay and increases treatment costs. Conventional treatments for respiratory muscles reverse these negative effects. İntensive care services are a set of services that have a very important place in public health care due to the vital support and they provide to all critically ill patients. This care services are constantly improving with the use of technological innovations. With the development of technology, virtual reality application has begun to be used therapeutically in the field of physiotherapy. Virtual reality is the combination of reality and imagination with fictions created using technology. Today, developers can surprisingly create realistic worlds filled with artificial intelligence that behaves believably. Studies have shown positive effects of virtual reality on acute respiratory frequency, pain and fatigue, and in light of this, it was predicted that it would be beneficial to apply to intensive care patients. This study will shed light on the rehabilitation of patients in intensive care and contribute to the literature.

DETAILED DESCRIPTION:
In the study, it was aimed to benefit from the effects of virtual reality application in intensive care patients and have a positive effect on vital signs and respiratory parameters in the early period.

This study will be randomly divided into two groups and it is planned to include 17 partipitants in each group. The first group will receive only conventional treatment, and the second group will receive virtual reality application in addition to conventional treatment. To evaluate the effectiveness of the application, vital signs, respiratory muscle strength, grip strength, blood gas analysis, shortness of breath and fatigue will be evaluated. Additionally, Richmond Agitation Sedation Scale (RASS), Nonverbal Pain Scale, Glaskow coma scale, Physical Function Test in Intensive Care (PFIT)-CPax (Chelsea Critical Care Physical Assessment Tool) scales will be used. All evaluations will be made before and after the application and a comparison will be made between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Individuals receiving inpatient treatment in intensive care who volunteer to participate in the research or who are allowed by their first-degree relatives if they are unconscious,
* Being over 18 years of age
* Being eligible to receive physiotherapy and rehabilitation from an intensive care physician
* Are in clinically stable condition

Exclusion Criteria:

* Patients with coagulation disorders (PT (Prothrombin Time); INR (International Normalized Ratio) value higher than 1.5 and platelet amount less than 50,000 m³)
* Patients with signs of increased intracranial pressure
* Skin wounds, ulcerations, allergic reactions
* Patients in contact isolation due to infection
* In shock
* Having malignancy
* Having multiple organ failure
* Having visual impairment
* Patients who are unconscious

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-06-08 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Respiratory Muscle Strength (MIP) | 3 days
  Maximal inspiratory pressure (MIP) is a measure of the strength of inspiratory muscles, primarily the diaphragm, and allows for the assessment of ventilatory failure, restrictive lung disease and respiratory muscle strength. MIP is measured at residual volume of lung.
Respiratory Muscle Strength (MEP) | 3 days
  For respiratory muscle strength, maximal expiratory pressure (MEP) will evaluate using an electronic pressure transducer. MEP is measured from total lung capacity.particularly the diaphragm, while MEPs measure the strength of abdominal and intercostal muscles.
  For respiratory muscle strength, maximal inspiratory pressure (MIP), and maximal expiratory pressure (MEP) were evaluated using an electronic pressure transducer. MIP was measured at residual volume, and MEP was measured from total lung capacity.
Richmond Agitation-Sedation Scale | 3 days
  Interrater reliability. In many intensive care units, the Richmond Agitation-Sedation Scale (RASS) is used to assess the level of sedation. This scale is designed with a three-step procedure that can help give a RASS score range of -5 to +4.The RASS score ranges from -5 (unarousable) to +4 (combative), with 0 meaning alert and calm.
SOFA (Sequential Organ Failure Assessment) | 3 days
  It evaluates morbidity through six systems (liver, central nervous system, respiratory system, cardiovascular system, renal and coagulation). For each system, points between 1 and 4 are given and the total score is evaluated between 6 and 24. In this score, as the score increases for each system, organ failure is considered to occur.
Visuel Anaolog Scale | 3 days
  A Visual Analogue Scale (VAS) is one of the pain rating scales used for the first time in 1921 by Hayes and Patterson[1]. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms.For pain intensity according to VAS, "no pain" is usually rated as 0 points and "worst pain imaginable" as 10 points. Ranges for pain intensity; <3. mild pain, 3-6 moderate pain, >6 severe pain
The Glasgow Coma Scale | 3 days
  It is a tool that healthcare providers use to measure decreases in consciousness. The scores from each section of the scale are useful for describing disruptions in nervous system function and also help providers track changes. It's the most widely used tool for measuring comas and decreases in consciousness.The components of the Glasgow Coma Scale include 4 different scores for the eye-opening response, 5 for the verbal response, and 6 for the motor response. The total score has values between 3 and 15. Three is the worst and 15 is the highest.
APACHE II Score | 3 days
  It is a general measure of disease severity based on current physiologic measurements, age & previous health conditions. The score can help in the assessment of patients to determine the level & degree of diagnostic & therapeutic intervention.APACHE II total score consists of three subheadings: acute physiology score, age and chronic health assessment; the highest value is 71. Mortality is 25% when the total score is 25, and increases to 80% when the total score is 35 and above.
Chelsea Critical Care Physical Assessment Tool (CPAx) | 3 days
  İt is a test used on male and female patients in the intensive care unit (ICU) to assess physical and respiratory function impairments and morbidity.
Body temperature | 3 days
  The average normal body temperature is generally accepted as 37°C. Some studies have shown that the "normal" body temperature can have a wide range, from 36.1°C to 37.2°C
Blood pressure | 3 days
  Normal blood pressure for most adults is defined as a systolic pressure of less than 120 and a diastolic pressure of less than 80. Elevated blood pressure is defined as a systolic pressure between 120 and 129 with a diastolic pressure of less than 80.
Respiratory rate | 3 days
  The normal range of breathing rate per minute in an average adult, for a person at rest, is 12 - 20 breaths per minute. Any person having a breathing rate under 12 or over 25 is considered to be breathing abnormally.
Pulse rate | 3 days
  The normal pulse for healthy adults ranges from 60 to 100 beats per minute. The pulse rate may fluctuate and increase with exercise, illness, injury, and emotions.
The Physical Function in ICU Test | 3 days
  The PFIT-s is a battery outcome measure involving four components: sit to stand assistance, marching on the spot cadence, shoulder flexor and knee extensor strength.

SECONDARY OUTCOMES:
Hand Strength | 3 days
  Hand muscle strength will be measured with a jamar device.
Modified Borg Dyspnea Scale | 3 days
  It is a categorical scale with a score from 0 to 10, where 0 represents normal breathing and 10 represents maximum dyspnea.
Pa02 | 3 days
  It is the partial pressure of oxygen in arterial blood. It is used to evaluate oxygenation. Normal values are 80-100 mmHg.
PaCO2 | 3 days
  It is the partial pressure of carbon dioxide in arterial blood. It is an indicator of alveolar ventilation. Normal values are 35-45 mmHg.
HCO3 | 3 days
  It is the serum concentration of bicarbonate ion. It is an important buffer in the blood and is used to evaluate the metabolic component of acid-base balance. Standard bicarbonate: It is the bicarbonate value that should be present in the blood under standard conditions (37°C temperature and 40 mmHg PCO2). Normally it is 22-26 mEq/L.
Ph | 3 days
  It is used to determine the H+ status of the blood. It shows that the patient is in acidosis or alkalosis, but it is not possible to understand the type by pH. Normal values are 7.35-7.45.
Confusion Assessment Method for the ICU | 3 days
  The Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) is a tool used to assess delirium among patients in the intensive care unit. The CAM-ICU assesses for the four features of delirium: Feature 1 is an acute change in mental status or a fluctuating mental status, Feature 2, is inattention, Feature 3, is altered level of consciousness and Feature 4, is disorganized thinking.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Çırak, Prof.Dr., Study Director — İstinye University
Locations (1):
- İstinye Üniversitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Study Protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF), Clinical Study Report (CSR) might be considered to be shared with clinicians studying in the same field one year after the publication of the study

REFERENCES:
- [Result] Berger D, Bloechlinger S, von Haehling S, Doehner W, Takala J, Z'Graggen WJ, Schefold JC. Dysfunction of respiratory muscles in critically ill patients on the intensive care unit. J Cachexia Sarcopenia Muscle. 2016 Sep;7(4):403-12. doi: 10.1002/jcsm.12108. Epub 2016 Mar 9. PMID 27030815
- [Result] Makhabah DN, Martino F, Ambrosino N. Peri-operative physiotherapy. Multidiscip Respir Med. 2013 Jan 23;8(1):4. doi: 10.1186/2049-6958-8-4. PMID 23343253
- [Result] Yousefnia-Darzi F, Hasavari F, Khaleghdoost T, Kazemnezhad-Leyli E, Khalili M. Effects of thoracic squeezing on airway secretion removal in mechanically ventilated patients. Iran J Nurs Midwifery Res. 2016 May-Jun;21(3):337-42. doi: 10.4103/1735-9066.180374. PMID 27186214
- [Result] Kalanuria AA, Ziai W, Mirski M. Ventilator-associated pneumonia in the ICU. Crit Care. 2014 Mar 18;18(2):208. doi: 10.1186/cc13775. No abstract available. PMID 25029020
- [Result] Ratnovsky A, Elad D, Halpern P. Mechanics of respiratory muscles. Respir Physiol Neurobiol. 2008 Nov 30;163(1-3):82-9. doi: 10.1016/j.resp.2008.04.019. Epub 2008 May 15. PMID 18583200
- [Result] Castro-Avila AC, Seron P, Fan E, Gaete M, Mickan S. Effect of Early Rehabilitation during Intensive Care Unit Stay on Functional Status: Systematic Review and Meta-Analysis. PLoS One. 2015 Jul 1;10(7):e0130722. doi: 10.1371/journal.pone.0130722. eCollection 2015. PMID 26132803
- [Result] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Result] Corner EJ, Wood H, Englebretsen C, Thomas A, Grant RL, Nikoletou D, Soni N. The Chelsea critical care physical assessment tool (CPAx): validation of an innovative new tool to measure physical morbidity in the general adult critical care population; an observational proof-of-concept pilot study. Physiotherapy. 2013 Mar;99(1):33-41. doi: 10.1016/j.physio.2012.01.003. Epub 2012 Mar 30. PMID 23219649
- [Result] Alves da Cruz MM, Ricci-Vitor AL, Bonini Borges GL, Fernanda da Silva P, Ribeiro F, Marques Vanderlei LC. Acute Hemodynamic Effects of Virtual Reality-Based Therapy in Patients of Cardiovascular Rehabilitation: A Cluster Randomized Crossover Trial. Arch Phys Med Rehabil. 2020 Apr;101(4):642-649. doi: 10.1016/j.apmr.2019.12.006. Epub 2020 Jan 8. PMID 31926142
- [Result] Taslimipour S, Rojhani-Shirazi Z, Hemmati L, Rezaei I. Effects of a Virtual Reality Dance Training Program on Kyphosis Angle and Respiratory Parameters in Young Women With Postural Hyperkyphosis: A Randomized Controlled Clinical Trial. J Sport Rehabil. 2020 May 13;30(2):293-299. doi: 10.1123/jsr.2019-0303. PMID 32404535
- [Result] Pazzaglia C, Imbimbo I, Tranchita E, Minganti C, Ricciardi D, Lo Monaco R, Parisi A, Padua L. Comparison of virtual reality rehabilitation and conventional rehabilitation in Parkinson's disease: a randomised controlled trial. Physiotherapy. 2020 Mar;106:36-42. doi: 10.1016/j.physio.2019.12.007. Epub 2019 Dec 23. PMID 32026844
- [Result] Rodrigues IM, Lima AG, Santos AED, Santos ACA, Nascimento LSD, Serra MVCL, Pereira TJS, Barbosa FDS, Seixas VM, Monte-Silva K, Scipioni KRDDS, Cruz DMCD, Piscitelli D, Goffredo M, Gois-Junior MB, Zanona AF. A Single Session of Virtual Reality Improved Tiredness, Shortness of Breath, Anxiety, Depression and Well-Being in Hospitalized Individuals with COVID-19: A Randomized Clinical Trial. J Pers Med. 2022 May 19;12(5):829. doi: 10.3390/jpm12050829. PMID 35629250
- [Result] Parker A, Sricharoenchai T, Needham DM. Early Rehabilitation in the Intensive Care Unit: Preventing Physical and Mental Health Impairments. Curr Phys Med Rehabil Rep. 2013 Dec;1(4):307-314. doi: 10.1007/s40141-013-0027-9. PMID 24436844
- [Result] Trampisch US, Franke J, Jedamzik N, Hinrichs T, Platen P. Optimal Jamar dynamometer handle position to assess maximal isometric hand grip strength in epidemiological studies. J Hand Surg Am. 2012 Nov;37(11):2368-73. doi: 10.1016/j.jhsa.2012.08.014. PMID 23101534
- [Result] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743